CLINICAL TRIAL: NCT05761600
Title: Group Art Therapy Practice for People With a Learning Disability (GATher-LD): A Qualitative Study
Brief Title: Learning Disability Group Art Therapy: Looking and Asking
Acronym: GATher-LD
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other); East London NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 147946
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Learning Disability, Adult; Mental Health
MeSH Terms: conditions — Learning Disabilities; Psychological Well-Being | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Art Therapist: Professionally qualified and HCPC registered Arts Therapists delivering group arts therapy in the community settings in the UK
  Interventions: Other: Ethnographically-informed group observation; Other: Semi-structured Interviews; Other: Focus Group
- People with a Learning Disability: Adults (18 years+) currently attending an art therapy group who have a learning disability and can consent and communicate in a way that supports meaningful engagement in the study.
  Interventions: Other: Ethnographically-informed group observation; Other: Semi-structured Interviews
- Identified Support Person: Person who is well-known to the person with a learning disability (e.g. NHS staff, paid support staff or family members who are carers) who provides practical and/or emotional support to the person with a learning disability attending the art therapy group
  Interventions: Other: Semi-structured Interviews

INTERVENTIONS:
Other: Ethnographically-informed group observation — The chief investigator will visit each art therapy group 3-6 times; there will be up to 5 groups recruited. They will record observational data and insights; making use of visual reflective journaling where appropriate. These will later be written up as full field notes.
  Groups: Art Therapist; People with a Learning Disability
Other: Semi-structured Interviews — Individual interviews will take place with all three key stakeholders in group art therapy at different stages of the study. Each interview will have a topic guide to structure the discussion and will combine arts-based methods with conversation to maximise accessibility. Interview location, timing and format (online or in-person) are flexible, and the chief investigator will adapt to the needs of the participants.
Other: Focus Group — After data collection and initial analysis (likely 3-5 months after final observation and/or interview) a focus group will be held with the art therapist participants. This session will use arts-based engagement to support member checking of the initial results and triangulation of the findings, which is likely to include potential active ingredients in group art therapy and principles of practice with this client group.
  Groups: Art Therapist

SUMMARY:
A qualitative study of group art therapy in England for adults with a learning disability accessing community services. Different stakeholder views and experiences will be gathered using ethnographically-informed group observation, semi-structured individual interviews and a focus group. People with a learning disability will support the data analysis and dissemination of findings in accessible means.

ELIGIBILITY:
INCLUSION CRITERIA:

Participants who are art therapists must:

* Be a HCPC registered arts therapist practicing in the UK
* Have experience of delivering group arts therapy in a community setting to this population
* Be able to give informed consent and communicate in English

Participants who are adults with a learning disability must:

* Be 18 years old or over
* Have a diagnosed learning disability or be accessing an NHS specialist learning disability service or using their personal budget to access a third sector art therapy group for this population
* Have experienced mental distress, have a diagnosed mental health condition or be accessing support for their mental health
* Be currently accessing group arts therapy
* Be able to give informed consent with adapted communication aids and approaches to meet their communication preferences
* Have a level of verbal ability to ensure they can communicate their views and meaningfully engage in the study

Participants who are paid support staff or family carers must:

* Be 18 years old or over
* Be identified by the person with a learning disability as someone who knows them well and could represent the carer perspective in this study
* Be able to give informed consent
* Have adequate command of the English to be able to meaningfully engage in the study

Participants will be excluded if they:

* Are unable to engage in the informed consent process; this is likely to exclude people who have a more severe form of learning disability
* Delivering the arts therapy group on an inpatient or acute ward
* Trainee arts therapists, or those who have yet to complete registration with the HCPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are three different participant groups in this study. They are:
  1. Professionally qualified and HCPC registered Arts Therapists delivering group arts therapy in the community settings in the UK
  2. Adults with a learning disability who are currently attending an arts therapy group
  3. An identified support person who is well-known to the service user (e.g. NHS staff, paid support staff or family members who are carers) who provides practical and/or emotional support to the person with a learning disability attending the art therapy group
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
To understand the features of current group art therapy practice for people with a learning disability | 12 months
  Through using ethnographically informed observation of art therapy groups, arts-based semi-structured interviews and focus group to gather key stakeholder perspectives from service users, carers, and art therapists

SECONDARY OUTCOMES:
Identify the potential active ingredients of art therapy with this client group through describing the procedures used by art therapists | 12 months
Understand how people with a learning disability experience art therapy to identify helpful therapist behaviours and highlight possible future domains of outcome measurement | 12 months
Identify the components of the intervention, which includes dynamic administration and how best to include the person's network | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicki Power, Principal Investigator — Queen Mary University of London
Locations (5):
- United Kingdom (5):
  - Oxleas NHS Foundation Trust, London, Kent
  - Northern Care Alliance NHS Foundation Trust, Salford, Manchester
  - Sirona Adult Learning Disability Health Service, Bristol
  - Coventry and Warwickshire NHS Foundation Trust, Coventry
  - East London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No